CLINICAL TRIAL: NCT00154986
Title: Study of IGFBP-3 in the Ovarian Carcinoma Cell Invasion
Brief Title: IGFBP-3 in Ovarian Cancer Invasion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 9361700500; NSC93-2314-B-002-168
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2005-09-12 (Estimated); Status verified 2004-04

CONDITIONS: Ovarian Carcinoma
Keywords: invasion; migration; metastasis; IGFBP-3; transfection; signal transduction.
MeSH Terms: conditions — Ovarian Neoplasms; Neoplasm Metastasis | interventions — Transfection

INTERVENTIONS:
Procedure: immunohistochemical staining, transfection, invasion assay

SUMMARY:
An ovarian cancer cell line (OVTW-59) derived from an ovarian endometrioid carcinoma was established and its sublines, labeled as P0, P1, P2, P3, and P4 with increasing invasion abilities were selected from transwell invasion chambers.Using cDNA microarray and verified with quantitative reverse-transcriptase polymerase chain reaction, we have identified IGFBP-3 as an invasion-suppressor gene. We plan to study the role of IGFBP-3 in ovarian cancer invasion.

DETAILED DESCRIPTION:
We have successfully established an ovarian cancer cell line (OVTW-59), which was derived from an ovarian endometrioid carcinoma. Its sublines, labeled as P0, P1, P2, P3, and P4 with increasing invasion abilities, were selected from transwell invasion chambers, where P0 represented the original cell line at 100th passage. By using cDNA microarray and verified with quantitative reverse-transcriptase polymerase chain reaction, we have identified the differentially gene expression profiles of these OVTW-59 series cell lines in order to identify the invasion related suppressor and oncogenes from ovarian carcinoma. From these genes, we selected insulin-like growth factor binding protein (IGFBP)-3, which is a suppressor gene, and found it lower expressed in higher-grade tumors and correlated with poor patient survival. In vitro, we found IGFBP-3 related to the inhibition of cancer cell migration. In this study, we plan to setup stable transfected IGFBP-3 cell lines in P0 and P4, and study the relationship among IGFBP-3, metalloproteinase-2 (our previous studies which verified its relationship with tumor invasiveness) and insulin-like growth factor (IGF)-1. We would study the changes in cytoskeletal structures and the known functions of anti-proliferation and apoptosis in IGFBP-3. Furthermore, we would like to investigate the mechanism of IGFBP-3 in the inhibition of invasion/migration of ovarian carcinoma, either signaling through MAPK or PI3K/AKT pathways. Finally, through xenograft, we plan to study for the possible application of IGFBP-3 in ovarian cancer therapy.

ELIGIBILITY:
Inclusion Criteria:

Ovarian Endometrioid Adenocarcinoma

Exclusion Criteria:

Other types of ovaria epithelial cell carcinoma

Ages: 21 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2004-08; Study Completion 2005-07

PRIMARY OUTCOMES:
migration, invasion, metastasis

SECONDARY OUTCOMES:
transfection efficiency

CONTACTS AND LOCATIONS:
Overall Officials: Torng Pao-Ling, MD, PhD, Principal Investigator — Department of Obsteteric and Gynecology, National Tiawan University Hospital
Locations (1):
- National Taiwna University Hospital, Taipei, Taiwan